CLINICAL TRIAL: NCT03849183
Title: The Effect of Subcutaneous Nitroglycerin on the Success Rate of Arterial Catheterization in Pediatric Patients: a Randomized Controlled Trial
Brief Title: Subcutaneous Nitroglycerin for Pediatric Radial Artery Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-1810-077-979
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Arterial Line
Keywords: Radial Artery; Vascular Catheters
MeSH Terms: interventions — Nitroglycerin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitroglycerin (Experimental): Nitroglycerin 5mcg/kg (0.5cc) is subcutaneously injected before radial artery cannulation.
  Interventions: Drug: Nitroglycerin
- Control (Active Comparator): Normal saline (0.5cc) is subcutaneously injected before radial artery cannulation.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Nitroglycerin — Subcutaneous nitroglycerin injection to increase the first attempt success rate of radial artery cannulation in pediatric patients
  Other Names: Subcutaneous Nitroglycerin
  Arms: Nitroglycerin
Drug: Normal saline — Subcutaneous normal saline injection to increase the first attempt success rate of radial artery cannulation in pediatric patients
  Other Names: Subcutaneous Normal saline
  Arms: Control

SUMMARY:
The primary objective of the study is to evaluate the vasodilative effect of subcutaneous nitroglycerin during ultrasound-guided radial artery cannulation in pediatric patients. The hypothesis of this study is that the subcutaneous nitroglycerin will increase the radial artery size and improve the first-attempt success rate of radial artery cannulation. This is a single-center, double-blind, randomized, placebo-controlled study comparing the effect of subcutaneous nitroglycerin and saline on radial artery cannulation in pediatric patients undergoing general anesthesia. Prior to the procedure, each patient will be randomized into either the control arm, saline, or study arm, nitroglycerin.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia
* Arterial cannulation for hemodynamic monitoring, multiple blood sample

Exclusion Criteria:

* Hypersensitivity or contraindication to nitroglycerine
* Unstable vital sign, significant arrhythmia or hypotension, Shock
* High risk of peripheral ischemia
* Skin disease, infection, hematoma, recent cannulation at radial artery.
* Increased intracranial pressure, Intracranial hemorrhage
* Glaucoma
* Recent use of PDE5 inhibitors (<24 hours after sildenafil or vardenafil; <48 hours after tadalafil)

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
First attempt success rate | During radial artery cannulation (up to 1 hour)
  Success at the first skin puncture

SECONDARY OUTCOMES:
Size of radial artery | Before and after subcutaneous injection of drugs (up to 1 hour)
  Internal diameter of radial artery
depth of radial artery | Before and after subcutaneous injection of drugs (up to 1 hour)
  depth of radial artery from the skin
Overall attempt | During radial artery cannulation (up to 1 hour)
  Number of attempt of radial artery cannulation
Overall Procedure time | During radial artery cannulation (up to 1 hour)
  From ultrasound guidance, to Arterial waveform
Overall success rate | During radial artery cannulation (up to 1 hour)
  Success within 4 skin puncture (2 skin puncture at each radial artery)
Malfunction of radial artery catheter | After radial artery cannulation assessed during anesthesia (up to 24 hour)
  Invasive blood pressure monitoring, Sampling
Complication rate | After radial artery cannulation assessed up to PACU, PICU stay (per 24hour, up to 48 hour)
  Hematoma, Distal ischemia, Spasm accessed by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chong AY, Lo T, George S, Ratib K, Mamas M, Nolan J. The effect of pre-procedure sublingual nitroglycerin on radial artery diameter and Allen's test outcome - Relevance to transradial catheterization. Cardiovasc Revasc Med. 2018 Mar;19(2):163-167. doi: 10.1016/j.carrev.2017.07.016. Epub 2017 Jul 29. PMID 28923695
- [Background] Chen Y, Ke Z, Xiao J, Lin M, Huang X, Yan C, Ye S, Tan X. Subcutaneous Injection of Nitroglycerin at the Radial Artery Puncture Site Reduces the Risk of Early Radial Artery Occlusion After Transradial Coronary Catheterization: A Randomized, Placebo-Controlled Clinical Trial. Circ Cardiovasc Interv. 2018 Jul;11(7):e006571. doi: 10.1161/CIRCINTERVENTIONS.118.006571. PMID 30002088
- [Background] Kim EH, Lee JH, Song IK, Kim JT, Lee WJ, Kim HS. Posterior Tibial Artery as an Alternative to the Radial Artery for Arterial Cannulation Site in Small Children: A Randomized Controlled Study. Anesthesiology. 2017 Sep;127(3):423-431. doi: 10.1097/ALN.0000000000001774. PMID 28682811
- [Background] Ezhumalai B, Satheesh S, Jayaraman B. Effects of subcutaneously infiltrated nitroglycerin on diameter, palpability, ease-of-puncture and pre-cannulation spasm of radial artery during transradial coronary angiography. Indian Heart J. 2014 Nov-Dec;66(6):593-7. doi: 10.1016/j.ihj.2014.05.023. Epub 2014 Jun 7. PMID 25634390
- [Background] Beyer AT, Ng R, Singh A, Zimmet J, Shunk K, Yeghiazarians Y, Ports TA, Boyle AJ. Topical nitroglycerin and lidocaine to dilate the radial artery prior to transradial cardiac catheterization: a randomized, placebo-controlled, double-blind clinical trial: the PRE-DILATE Study. Int J Cardiol. 2013 Oct 3;168(3):2575-8. doi: 10.1016/j.ijcard.2013.03.048. Epub 2013 Apr 10. PMID 23582415
- [Background] Majure DT, Hallaux M, Yeghiazarians Y, Boyle AJ. Topical nitroglycerin and lidocaine locally vasodilate the radial artery without affecting systemic blood pressure: a dose-finding phase I study. J Crit Care. 2012 Oct;27(5):532.e9-13. doi: 10.1016/j.jcrc.2012.04.019. Epub 2012 Jun 12. PMID 22699036